CLINICAL TRIAL: NCT06529068
Title: Blood Pressure Responses to Isometric Blood Flow Restriction Exercise
Brief Title: Cardiovascular Response to Isometric BFR Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00006378
Record Dates: First submitted 2024-07-18; First posted 2024-07-31 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isometric exercise without BFR cuff (control) (Active Comparator)
  Interventions: Behavioral: Isometric handgrip exercise
- Isometric exercise with narrow-elastic BFR band (Experimental)
  Interventions: Behavioral: Isometric handgrip exercise with a narrow-elastic band
- Isometric exercise with wide-rigid BFR cuff (Experimental)
  Interventions: Behavioral: Isometric handgrip exercise with a wide-rigid cuff

INTERVENTIONS:
Behavioral: Isometric handgrip exercise — The participants will perform isometric handgrip exercises without blood flow restriction.
  Arms: Isometric exercise without BFR cuff (control)
Behavioral: Isometric handgrip exercise with a narrow-elastic band — The participants will perform isometric handgrip exercises with blood flow restriction using a narrow-elastic band.
  Arms: Isometric exercise with narrow-elastic BFR band
Behavioral: Isometric handgrip exercise with a wide-rigid cuff — The participants will perform isometric handgrip exercises with blood flow restriction using a wide-rigid cuff.
  Arms: Isometric exercise with wide-rigid BFR cuff

SUMMARY:
The goal of this interventional study is to evaluate the acute impact of isometric blood flow restriction (BFR) exercise on blood pressure and other cardiovascular functions in healthy young adult volunteers. The main question it aims to answer is:

The investigators hypothesize that isometric BFR exercise with a wide-rigid cuff would lead to greater blood pressure and other cardiovascular responses and that these cardiovascular responses would be greater under isometric BFR exercise with narrow-elastic bands compared with the control condition (no cuff).

Participants will perform isometric exercises in 3 laboratory visits with different exercise conditions) no cuff control 2) BFR with wide-rigid cuff 3) BFR with narrow-elastic band.

ELIGIBILITY:
Inclusion Criteria:

- Apparently healthy young adults aged between 18 - 40 years old and signed the informed consent.

Exclusion Criteria:

* Abnormal clotting times
* Acid-base imbalance/acidosis
* Arterial calcification
* Atherosclerotic vessels
* Cardiopulmonary conditions
* Diabetes
* Dialysis/central venous access
* General/local infection
* High intracranial pressure
* Hip, pelvis, or femur fracture
* History of venous thromboembolism
* Hypertension
* Immobility for greater than 48 hours in the past month
* Immobilizing cast
* Implanted medical device
* Lymphectomies
* Obesity
* Open fracture
* Open or unhealed soft tissue injuries
* Paralysis
* Peripheral vascular disease
* Pregnancy/postpartum
* Prior revascularization
* Renal compromise
* Severe crush injuries
* Sickle cell trait/anemia
* Skin grafts
* Stroke
* Temporary nerve damage
* Thrombophilia
* Tumor/cancer
* Varicose veins
* Vascular grafting

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure and diastolic blood pressure | 20 minutes
  Beat-by-beat (both systolic and diastolic blood pressure) blood pressure before, during, and after exercise
Brachial artery diameter evaluated by an ultrasound machine | Before and 20 minutes after exercise
  Brachial artery diameter will be measured by an ultrasound machine to calculate flow-mediated dilation (FMD)
Heart rate | 20 minutes
  Monitor heart rate continuously before, during, and after exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Aging Research Laboratory, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lind AR. Cardiovascular responses to static exercise. (Isometrics, anyone?). Circulation. 1970 Feb;41(2):173-6. doi: 10.1161/01.cir.41.2.173. No abstract available. PMID 5412979
- [Background] Domingos E, Polito MD. Blood pressure response between resistance exercise with and without blood flow restriction: A systematic review and meta-analysis. Life Sci. 2018 Sep 15;209:122-131. doi: 10.1016/j.lfs.2018.08.006. Epub 2018 Aug 4. PMID 30086274
- [Background] Bond CW, Hackney KJ, Brown SL, Noonan BC. Blood Flow Restriction Resistance Exercise as a Rehabilitation Modality Following Orthopaedic Surgery: A Review of Venous Thromboembolism Risk. J Orthop Sports Phys Ther. 2019 Jan;49(1):17-27. doi: 10.2519/jospt.2019.8375. Epub 2018 Sep 12. PMID 30208794
- [Background] Mannozzi J, Al-Hassan MH, Kaur J, Lessanework B, Alvarez A, Massoud L, Aoun K, Spranger M, O'Leary DS. Blood flow restriction training activates the muscle metaboreflex during low-intensity sustained exercise. J Appl Physiol (1985). 2023 Aug 1;135(2):260-270. doi: 10.1152/japplphysiol.00274.2023. Epub 2023 Jun 22. PMID 37348015
- [Background] Song JS, Yamada Y, Wong V, Bell ZW, Spitz RW, Abe T, Loenneke JP. Hypoalgesia following isometric handgrip exercise with and without blood flow restriction is not mediated by discomfort nor changes in systolic blood pressure. J Sports Sci. 2022 Mar;40(5):518-526. doi: 10.1080/02640414.2021.2003569. Epub 2021 Nov 25. PMID 34823439
- [Background] Renzi CP, Tanaka H, Sugawara J. Effects of leg blood flow restriction during walking on cardiovascular function. Med Sci Sports Exerc. 2010 Apr;42(4):726-32. doi: 10.1249/MSS.0b013e3181bdb454. PMID 19952840
- [Background] Early KS, Rockhill M, Bryan A, Tyo B, Buuck D, McGinty J. EFFECT OF BLOOD FLOW RESTRICTION TRAINING ON MUSCULAR PERFORMANCE, PAIN AND VASCULAR FUNCTION. Int J Sports Phys Ther. 2020 Dec;15(6):892-900. doi: 10.26603/ijspt20200892. PMID 33344005
- [Background] Credeur DP, Hollis BC, Welsch MA. Effects of handgrip training with venous restriction on brachial artery vasodilation. Med Sci Sports Exerc. 2010 Jul;42(7):1296-302. doi: 10.1249/MSS.0b013e3181ca7b06. PMID 20019641
- [Background] Schneider AC, Hughes WE, Ueda K, Bock JM, Casey DP. Reduced blood pressure responsiveness to skeletal muscle metaboreflex activation in older adults following inorganic nitrate supplementation. Nitric Oxide. 2018 Aug 1;78:81-88. doi: 10.1016/j.niox.2018.05.010. Epub 2018 Jun 1. PMID 29864505